CLINICAL TRIAL: NCT03695484
Title: Prospective, Multicenter, Non-randomized Observational Registry Conducted at High Volume Experienced Treatment Centers Utilizing the Most Current AF Ablation Techniques.
Brief Title: Registry Evaluating AF Ablation Techniques
Acronym: PRIME-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Anne-Marie Noten, Principal investigator, Erasmus Medical Center
Other Study IDs: PRIME-AF
Record Dates: First submitted 2018-09-20; First posted 2018-10-04 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation; Catheter Ablation
Keywords: Paroxysmal Atrial Fibrillation; Catheter Ablation; Cryoballoon; Radiofrequency ablation; Remote Magnetic Navigation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Manual guided RF ablation: Patients with paroxysmal atrial fibrillation treated with Manual guided RF ablation using Contact Force catheters
- Cryoballoon ablation: Patients with paroxysmal atrial fibrillation treated with Cryoballoon ablation. Cryoballoon: Arctic Front Advance, Medtronic - 28 mm
- RMN guided RF ablation - High power: Patients with paroxysmal atrial fibrillation treated with Remote Magnetic Navigation guided RF ablation with e-Contact and high power settings.
  High power ablation settings: a minimum of 40 Watt, 43grC, flow 17ml/min. Higher voltages (e.g. anterior wall) are allowed with respect to the operators' preference.
- RMN guided RF ablation - Low power: Patients with paroxysmal atrial fibrillation treated with Remote Magnetic Navigation guided RF ablation with e-Contact and low power settings.
  Low power ablation settings: a maximum of 39 Watt, 43grC, flow 17ml/min. Lower voltages are allowed with respect to the operators' preference.

SUMMARY:
The purpose of this observational registry is to prospectively collect procedure efficiency, safety and acute and long term outcome data from catheter ablation procedures as treatment of paroxysmal atrial fibrillation, using the following treatment modalities:

* Cryoballoon ablation
* Manual guided RF ablation using Contact Force catheters
* Remote Magnetic Navigation guided RF ablation with e-Contact and high power settings
* Remote Magnetic Navigation guided RF ablation with e-Contact and low power settings

ELIGIBILITY:
Inclusion Criteria:

* Documented Paroxysmal Atrial Fibrillation
* Eligibility for Pulmonary Vein Isolation by catheter ablation based on the respective ACC/AHA/ESC Guideline valid at the date of procedure
* Signed the informed consent to participate in the registry

Exclusion Criteria:

* Younger than 18 years of age
* Prior AF ablation procedure (including MAZE procedure)
* Prior ablation of Non-AF Arrhythmia within 3 months of enrollment
* Presence of cardiac thrombus
* Other AF ablations performed during procedure (e.g. lines, rotor, CFAE's etc)
* Active endocarditis or systemic infection
* Life expectancy < 1 year
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for participation in the study have a reported incidence of at least two documented episodes of symptomatic paroxysmal atrial fibrillation during the three months preceding trial entry, as well as documentation of at least one episode of AF on ECG, and are eligible for PVI by catheter ablation based on the respective ACC/AHA/ESC Guideline valid at the date of procedure
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Procedure time | During ablation procedure
  Procedure time (minutes)
Fluoroscopy time | During ablation procedure
  Fluoroscopy time (minutes)
Transseptal time | During ablation procedure
  Transseptal time (time from insertion of catheters until transseptal puncture) (minutes)
Left atrial dwell time | During ablation procedure
  Left atrial dwell time (time from LA entry until removal of catheters) (minutes)
PVI ablation time | During ablation procedure
  PVI ablation time (total PVI ablation time, i.e. first until last application) (minutes)
Ablation time per pulmonary vein | During ablation procedure
  Ablation time per pulmonary vein (minutes)

SECONDARY OUTCOMES:
First Pass Isolation | During ablation procedure
  First Pass Isolation (i.e. Successful isolation of PVs after the first ablation attempt)
Acute success | During ablation procedure
  Acute success (Successful electrical isolation of PVs at the end of procedure)
TouchUp rates | During ablation procedure
  TouchUp rates (additional applications for successful PV isolation)
Long-term success | From the date of procedure until 1 year
  Long-term success (freedom of atrial fibrillation 12 months after ablation)
Procedure-related adverse-events | From the date of procedure until 7 days
  Procedure-related adverse-events
Long-term adverse events | From the date of procedure until 1 year
  Long-term adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- Ziekenhuis Netwerk Antwerpen, Antwerp, Belgium
- Erasmus MC, Rotterdam, Netherlands
- E. Meshalkin National medical research center, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No